CLINICAL TRIAL: NCT00715351
Title: Efficacy and Safety of Glycaemic Control of Levemir® or Insulatard® in Patients With Type 2 Diabetes
Brief Title: Observational Study of Patients Using Levemir® or Insulatard® as Start Insulin for Treatment of Diabetes
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN304-1896
Record Dates: First submitted 2008-07-11; First posted 2008-07-15 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir; Insulin, Isophane

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- A
  Interventions: Drug: insulin detemir
- B
  Interventions: Drug: insulin NPH

INTERVENTIONS:
Drug: insulin detemir — Physician decides which insulin should be prescribed, selection of subjects will be at the discretion of participating physician
  Groups: A
Drug: insulin NPH — Physician decides which insulin should be prescribed, selection of subjects will be at the discretion of participating physician
  Groups: B

SUMMARY:
This trial is conducted in Europe. The aim of this observational study is to evaluate the glycaemic control, weight change and hypoglycaemic effects in patients with type 2 diabetes with Levemir® compared to Insulatard® under normal clinical practice conditions.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes failing on oral blood glucose lowering therapy, and requiring insulin therapy.

Exclusion Criteria:

* Type 1 diabetes
* Previous use of insulin

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Insulin naïve patients with type 2 diabetes treated with oral antidiabetics
Sampling Method: Non-Probability Sample
Enrollment: 342 (Actual)
Dates: Start 2007-05; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Body weight change | at 3 months and 6 months after baseline

SECONDARY OUTCOMES:
Hypoglycemic events | at 3 months and 6 months after baseline
Changes in glycaemic parameters | at 3 months and 6 months after baseline
Safety parameters by collecting (serious) adverse events and the pregnancies. | at 3 months and 6 months after baseline
Evaluation of general well-being by using the WHO-5 well-being questionnaire (Appendix I). | at 3 months and 6 months after baseline
Treatment satisfaction of subjects treated with insulin Levemir or NPH insulin by using insulin satisfaction ('Tevredenheid met insuline behandeling': Appendix II) | at 3 months and 6 months after baseline
Satisfaction of physicians who treat the subjects with insulin Levemir or NPH in-sulin by using a scale of 0-10 (Appendix III). | at 3 months and 6 months after baseline
Changes in doses | at 3 months and 6 months after baseline
HbA1c | at 3 months and 6 months after baseline
Changes in daily blood glucose values | at 3 months and 6 months after baseline

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Ljubljana, Slovenia

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com